CLINICAL TRIAL: NCT05977452
Title: The Risk Assessment Scale for Peripherally Inserted Central Venous Catheter (PICC) Related Thrombosis in Cancer Patients :A Prospective Study
Brief Title: The Risk Assessment Scale for Peripherally Inserted Central Venous Catheter (PICC) Related Thrombosis in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zeyin Hu, Infusion Therapy Specialist Nurse, Sun Yat-sen University
Other Study IDs: SunYat-senU 7-18
Record Dates: First submitted 2023-07-18; First posted 2023-08-04 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Thrombosis; Catheter
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with PICC placement
  Interventions: Diagnostic Test: Michigan Risk Score, Caprini Risk Assessment Model , Maneval scale

INTERVENTIONS:
Diagnostic Test: Michigan Risk Score, Caprini Risk Assessment Model , Maneval scale — Patients with PICC placement will be assessed by the Michigan Risk Score, Caprini Risk Assessment Model , Maneval scale（Chinese version） to predict the risk of PICC-related thrombosis. The time of evaluation are the day during PICC placement, 24-48h after PICC placement, and every time when patients receive PICC maintenance.

SUMMARY:
The aim of this study is to compare the accuracy and clinical predictive value of the Michigan Risk Score, Caprini Risk Assessment Model , and Maneval Scale （Chinese version）in predicting PICC-related thrombosis.

DETAILED DESCRIPTION:
The aim of this study is to compare the accuracy and clinical predictive value of the Michigan Risk Score, Caprini Risk Assessment Model , and Maneval Scale（Chinese version） in predicting PICC-related thrombosis.

Patients who will receive PICC placement will be evaluated by using the Michigan Risk Score, Caprini Risk Assessment Model , and Maneval Scale the day during PICC placement, 24-48h after PICC placement and every time patients receive PICC maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients
* Older than 18 years
* Being able to complete the questionnaire independently
* Patients who need PICC for treatment
* Being able to perform catheter maintenance in the hospital of admission until catheter removal
* Patients who agree to participate and sign the consent form

Exclusion Criteria:

* Patients who were or suspected to be allergic to the ingredients contained in PICC
* PICC placed in the lower extremity

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: cancer patients with PICC placement in Sun Yat-sen University Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
PICC thrombosis | through study completion，up to 1 year
  symptomatic thrombosis，diagnosed by symptoms such as pain, tenderness and swelling of the affected part and the verification of color doppler ultrasound of venous vessels
The Michigan Risk Score | From date of PICC catheterization until the date of PICC removal or date of occurrence of PICC related thrombosis, whichever came first, assessed up to 12 months.
  The risk score will be assessed. In this scale，risk factors associated with PICC-DVT included: history of DVT; multi-lumen PICC; active cancer; presence of another CVC when the PICC was placed; and white blood cell count greater than 12 000. The total score on the scale are 0 to 14 points, with a higher score indicates higher risk of thrombosis.
Maneval Scale | From date of PICC catheterization until the date of PICC removal or date of occurrence of PICC related thrombosis, whichever came first, assessed up to 12 months.
  The risk score will be assessed. This scale includes 45 risk factors associated with PICC thrombosis. The total score on the scale are 0 to 45 points, with a higher score indicates higher risk of thrombosis.
Caprini Risk Assessment Model | From date of PICC catheterization until the date of PICC removal or date of occurrence of PICC related thrombosis, whichever came first, assessed up to 12 months.
  The risk score will be assessed. This scale includes more than 40 risk factors associated with PICC thrombosis. In this scale，a higher score indicates higher risk of thrombosis.

CONTACTS AND LOCATIONS:
Locations (1):
- The Catheter Clinic, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided